CLINICAL TRIAL: NCT06617065
Title: A Prospective, Open-label Self-controlled Trial to Assess Long-term Changes in Pain and Function with Addition of 5% Dextrose to Local Anesthetic Solutions - the PALPADE Study
Brief Title: Exploring Long-term Pain Relief with 5% Dextrose Added to Local Anesthetic
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Seekers Centre (Other)
Responsible Party: Principal Investigator, Richard Nahas, Physician/Clinic director/ Principal investigator, The Seekers Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11997-RNahas
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-09

CONDITIONS: Chronic Non-cancer Pain
Keywords: Dextrose; Local anesthetics; Prolotherapy; Chronic pain; Interventional pain treatment; Peripheral nerve block
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Addition of 1 mL of 50% dextrose solution to the usual local anesthetic solution of choice (Experimental): The physician will add 1 mL of 50% dextrose solution (Pfizer Canada ULS, Kirkland, Québec) to the usual local anesthetic solution of choice for each patient. Solutions contain either 0.3% Ropivacaine, 1% Procaine, 0.5% Lidocaine, 0.25% Bupivacaine, or a mixture of 0.25% Bupivacaine and 2% Lidocaine in a 9:1 ratio.
  Interventions: Drug: Addition of 1 mL of 50% dextrose solution to the usual local anesthetic solution of choice for each patient.

INTERVENTIONS:
Drug: Addition of 1 mL of 50% dextrose solution to the usual local anesthetic solution of choice for each patient. — The principal investigator will use a palpation-guided approach to select the injection sites. Injection solutions will be prepared by the assisting nurse. For each patient, 1 mL of a 50% dextrose solution (Pfizer Canada ULS, Kirkland, Québec) will be added to the usual local anesthetic solution of choice.
  Solutions contain either 0.3% Ropivacaine, 1% Procaine, 0.5% Lidocaine, 0.25% Bupivacaine, or a mixture of 0.25% Bupivacaine and 2% Lidocaine in a 9:1 ratio.

SUMMARY:
The goal of this single-arm, non-randomized, open-label trial is to determine whether adding a 5% dextrose solution to a local anesthetic can improve outcomes in patients with chronic non-cancer pain.

The main question we aim to answer is whether adding a low-concentration (5%) dextrose solution to local anesthetics increases the effectiveness of trigger point injections and/or peripheral nerve blockade in the treatment of chronic non-cancer pain.

Researchers will compare the outcomes of adding 5% dextrose to the usual local anesthetic solution with the outcomes of using the local anesthetic alone to determine if injection therapy is more effective when dextrose is added.

Participants will:

* Attend their scheduled injection treatments every two (2) weeks for a total of six (6) visits.
* Complete a demographic form at the first visit, and the usual pre-visit questionnaires (the Waiting Room Form and the Brief Pain Inventory (BPI)) at every visit, as well as four (4) weeks after the sixth visit (approximately 16 weeks from the study start date). They will also need to complete two short questionnaires-the Patient Health Questionnaire (PHQ-9) and the Patient Global Impression of Change (PGIC)-at the specified intervals.
* Complete all forms, which will be securely emailed to them.

DETAILED DESCRIPTION:
Study Background:

There are many different approaches to treating chronic non-cancer pain, offering potential benefits such as symptom reduction, improved function, and enhanced quality of life. In most cases, conservative and noninvasive treatments are used first, with interventional procedures pursued for more persistent, severe, or disabling symptoms, either for diagnosis or treatment.

Injection treatments are typically considered when functional limitations persist despite physiotherapy, pharmacotherapy, and other non-invasive treatments. Corticosteroid injections into spinal and non-spinal joints, tendons, and ligaments are widely used, but repeated use has been associated with cartilage damage and tissue atrophy. Consequently, there is growing interest in other injectable solutions with potential benefits in pain management, including local anesthetics, dextrose, and platelet-rich plasma (PRP).

Prolotherapy is a non-surgical regenerative injection technique in which dextrose is delivered to tissues with degenerative damage, such as tendon insertions (entheses), joints, ligaments, and surrounding joint spaces. These injections are administered in a series of procedures at regular intervals. While the precise mechanism of action for prolotherapy remains unclear, some evidence suggests that a localized inflammatory cascade leads to collagen deposition and the release of growth factors. The increasing interest in prolotherapy is supported by a growing number of published intervention studies, which back anecdotal reports of its benefits in several painful conditions, with minimal adverse effects.

Dextrose has also been used as a diluent for local anesthetics, as it is soluble and does not cause pain or residual complications over time. Faiz et al. demonstrated that the addition of 5% dextrose to 0.5% bupivacaine provided an earlier onset of sensory block for the median nerve compared to normal saline. Additionally, Topol et al. showed superior effects of 1% lidocaine with 12.5% dextrose over lidocaine alone in adolescents with Osgood-Schlatter disease. While dextrose prolotherapy has been studied in several localized pain conditions, there is a lack of data on its role in generalized myofascial pain.

Our community-based pain clinic has been using repeated injections of local anesthetics as maintenance therapy for patients with chronic non-cancer pain. The purpose of this study is to assess the potential for dextrose to improve outcomes in these patients by delivering their usual local anesthetic in a 5% dextrose solution. Patients will receive six treatments over approximately three months, with long-term improvement measured by comparing outcomes at baseline, at the end of treatment, and four weeks after the final treatment, following the IMMPACT guidelines that inform this study's methodology.

This study is significant because it will be the first to compare the outcomes of injection treatment using local anesthetics with dextrose to local anesthetics alone, using a low concentration of dextrose, in a series of treatments to identify long-term improvements in chronic non-cancer pain. The hypothesis is that injection therapy will be more effective when dextrose is added, supporting the recommendation that dextrose should be routinely included in local anesthetic solutions for injection-based pain treatments. Our research question aims to determine whether adding a low-concentration (5%) dextrose solution to local anesthetics increases the effectiveness of trigger point injections and/or peripheral nerve blockade in the treatment of chronic non-cancer pain.

METHODS and MATERIALS

Study Design:

This study will be a single-arm, non-randomized, open-label trial. Patients with chronic non-cancer pain who are currently receiving routine care at a community-based pain clinic will be invited to participate. Eligible patients must have been receiving peripheral nerve blocks and trigger point injections for the management of their chronic pain for at least six months prior to enrollment. A 50% dextrose solution will be used to achieve a final concentration of 5% dextrose in addition to their usual local anesthetic solution. The results will be compared with historical data from when they received only nerve blocks.

DATA COLLECTION

Patient Demographics:

Demographic information will be collected, including age, gender, BMI, duration of symptoms, employment status, and pain intensity (measured using a Visual Analogue Scale). Additionally, during the initial visit, nurses will conduct a clinical assessment to determine the primary diagnosis, review current medications, and screen for mental illness, cognitive impairment, comorbidities, and prior spinal surgery.

Intervention:

The Principal Investigator will use a palpation-guided approach to choose injection sites. Injection solutions will be prepared by clinic nurses. 1 mL of 50% dextrose solution (Pfizer Canada ULS, Kirkland, Québec) will be added to the usual local anesthetic solution of choice for each patient. Solutions contain either 0.3% Ropivacaine, 1% Procaine, 0.5% Lidocaine, 0.25% Bupivacaine, or a mixture of 0.25% Bupivacaine and 2% Lidocaine in a 9:1 ratio.

The palpation-guided injection technique uses a novel approach to identify hypersensitive sensory fibres associated with pain generators in myofascial tissues and related structures. The procedure involves lightly sliding the fingertips along the skin in a linear direction (approximately 2-3 centimetres per second) until a palpable stress response is detected, which can be described as a change in skin turgor or tissue tension that can be felt by the examiner. This subtle but clearly discernible response may represent a lower threshold activation of the nociceptive flexion reflex (NFR), a widely used marker of central sensitization. Efforts are underway to evaluate the reliability of this palpation technique and its potential as a reliable, noninvasive tool for evaluating and treating painful disorders. Patients will receive this intervention a total of six times every 1-3 weeks, following their usual injection treatment schedule.

Clinical Measures:

Intervention data and patient-reported outcomes data will be extracted from routinely collected data, using the OceanMD platform. Patient-reported outcomes data will include the Brief Pain Inventory form (BPI), Patient Health Questionnaire (PHQ-9), duration of pain relief, and pain on a Visual Analogue Scale (VAS) ranging from 0 to 10 at the first visit (baseline/week 1), the third visit (week 5), the sixth and final visit (end of the intervention period/week 11), and again four weeks after the end of the intervention period (week 15). In addition, the Patient's Global Impression of the Change (PGIC) will also be measured at the end of the intervention (week 11) and four weeks later (week 15). Intervention data will include the number of injections, injection sites, and local anesthetic solutions used. Moreover, patients will fill out the usual waiting room questionnaire at every visit.

Rescue Treatment:

Patients who require urgent care for an acute injury or pain flare will be assessed and treated following usual protocols. Rescue injections and any other treatment administered will be based solely on the physician's judgment and will be documented in the patient's usual clinical chart notes (OSCAR EMR version 15).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years old, inclusive.
2. A primary diagnosis of chronic non-cancer pain as determined by their physician.
3. Present chronic pain symptoms of at least 3 months in duration.
4. Currently receiving injection therapy every 1-3 weeks for at least 6 months.
5. English proficiency

Exclusion Criteria:

1. Age less than 18 years
2. Scar or infection at the blockade puncture site
3. Pregnancy
4. Unstable neurologic or psychiatric diagnosis, including schizophrenia, bipolar disorder, substance use disorder, depression or anxiety, dementia or neurodegenerative disorder
5. Serious acute life stressor, clinical illness, or organ disease within the past three months
6. Serious or significant traumatic injury, surgical or dental procedure within the past three months
7. Lack of English proficiency or unable to complete patient forms
8. Denial or withdrawal of consent, as per the informed consent form (ICF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory form (BPI) | BPI is administered at the following intervals: first visit (Baseline/week 1), the third visit (Week 5), the sixth and final visit (Week 11), and again four weeks after the end of the intervention period (Week 15).
  The BPI allows patients to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function.
Patient Health Questionnaire (PHQ-9) | The PHQ-9 is administered at the following intervals: At the first visit (Baseline/Week 1), the third visit (Week 5), the sixth and final visit (Week 11), and again four weeks after the end of the intervention period (Week 15).
  The PHQ-9 is a depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
Visual Analogue Scale (VAS) | The VAS is administered at the following intervals: At the first visit (Baseline/Week 1), the third visit (Week 5), the sixth and final visit (Week 11), and again four weeks after the end of the intervention period (Week 15).
  VAS consists of a 10 cm horizontal line with the endpoints defining extreme limits such as no pain at all and pain as bad as possible.
Patient's Global Impression of the Change (PGIC) | The PGIC is administered at the following intervals: At the end of the intervention (Week 11) and four weeks after the end of the intervention period (Week 15).
  The PGIC is a short questionnaire that provides a responsive and interpretable assessment of how a participant evaluates changes in their status.

CONTACTS AND LOCATIONS:
Locations (1):
- Seekers Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected and stored using tablet-based case report forms on the PIPHA-compliant OCEAN platform (Well Health Technologies, Canada). All data will be anonymized, with direct identifiers removed and replaced by a unique study ID code.
  The study protocol, anonymized participant outcome data, and related data analysis will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: The IPD will be made available to approved researchers 12 months after the publication of the main study results. This period allows sufficient time for meticulous data preparation for external use.
Access Criteria: Access to IPD will be granted to researchers who submit scientifically valid proposals that align with ethical guidelines. A review committee will evaluate proposals based on their objectives, methodology, and compliance with data protection standards. Successful applicants will be required to sign a data use agreement outlining secure data handling and confidentiality requirements. Instructions for secure data access, including anonymization protocols and secure transfer methods, will be provided to approved researchers.

REFERENCES:
- [Background] Patel KV, Amtmann D, Jensen MP, Smith SM, Veasley C, Turk DC. Clinical outcome assessment in clinical trials of chronic pain treatments. Pain Rep. 2021 Jan 21;6(1):e784. doi: 10.1097/PR9.0000000000000784. eCollection 2021 Jan-Feb. PMID 33521482
- [Background] Bae G, Kim S, Lee S, Lee WY, Lim Y. Prolotherapy for the patients with chronic musculoskeletal pain: systematic review and meta-analysis. Anesth Pain Med (Seoul). 2021 Jan;16(1):81-95. doi: 10.17085/apm.20078. Epub 2020 Dec 16. PMID 33348947
- [Background] Hauser RA, Lackner JB, Steilen-Matias D, Harris DK. A Systematic Review of Dextrose Prolotherapy for Chronic Musculoskeletal Pain. Clin Med Insights Arthritis Musculoskelet Disord. 2016 Jul 7;9:139-59. doi: 10.4137/CMAMD.S39160. eCollection 2016. PMID 27429562
- [Background] Wee TC, Neo EJR, Tan YL. Dextrose prolotherapy in knee osteoarthritis: A systematic review and meta-analysis. J Clin Orthop Trauma. 2021 May 20;19:108-117. doi: 10.1016/j.jcot.2021.05.015. eCollection 2021 Aug. PMID 34046305
- [Background] Rabago D, Slattengren A, Zgierska A. Prolotherapy in primary care practice. Prim Care. 2010 Mar;37(1):65-80. doi: 10.1016/j.pop.2009.09.013. PMID 20188998
- [Background] Hung CY, Hsiao MY, Chang KV, Han DS, Wang TG. Comparative effectiveness of dextrose prolotherapy versus control injections and exercise in the management of osteoarthritis pain: a systematic review and meta-analysis. J Pain Res. 2016 Oct 18;9:847-857. doi: 10.2147/JPR.S118669. eCollection 2016. PMID 27799816
- [Background] Goswami A. Prolotherapy. J Pain Palliat Care Pharmacother. 2012 Dec;26(4):376-8. doi: 10.3109/15360288.2012.734900. PMID 23216178